CLINICAL TRIAL: NCT01727063
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy of Intramyocardial Injection of Autologous Bone-Marrow Cells in Patients With Severe, Chronic Ischemic Heart Disease Undergoing Coronary Bypass Surgery
Brief Title: Cell Therapy in Severe Chronic Ischemic Heart Disease
Acronym: MiHeart
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Luis Henrique W Gowdak, MD, PhD, Clinical Coordinator, Ministry of Health, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMRTCC-ISQ2
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Chronic Ischemic Heart Disease; Coronary Artery Disease; Angina Pectoris
Keywords: Chronic ischemic heart disease; Coronary artery disease; Angina pectoris; Myocardial ischemia; Cardiac surgery
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Ischemia | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Intervention Model Description: Intramyocardial injection of bone marrow-derived cells OR placebo (saline) during CABG
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cell Therapy (Experimental): Intramyocardial injection of autologous bone marrow-derived cells
  Interventions: Procedure: Cell Therapy
- Placebo (No Intervention): Saline injection

INTERVENTIONS:
Procedure: Cell Therapy — Intramyocardial injection of autologous bone marrow-derived cells
  Arms: Cell Therapy

SUMMARY:
Patients with advanced coronary artery disease usually undergo incomplete myocardial revascularization due to the extension and diffuseness of the disease, with very poor distal arterial beds unsuitable for direct revascularization.

This study was designed to test the hypothesis that direct, intramyocardial injection of autologous bone marrow cells may further improve myocardial perfusion in patients undergoing incomplete bypass surgery.

DETAILED DESCRIPTION:
All eligible patients will undergo coronary artery bypass grafting (CABG) and, in previously identified areas of viable, ischemic myocardium unsuitable for direct revascularization, be randomized to either placebo (saline) or intramyocardial injection of bone marrow-derived cells (BMC) during surgery.

During follow-up, myocardial perfusion assessment will be performed to determine the improvement in treated areas compared to non-treated segments.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of angina or angina equivalent
* documented coronary artery disease (invasive angiography)
* documented myocardial ischemia (stress echo, cardiac scintigraphy, or MRI)
* unsuitable for complete myocardial revascularization (PCI or CABG) OR even if a complete procedure in feasible, it is anticipated that myocardial perfusion may not be restored due to poor distal beds

Exclusion Criteria:

* severe LV dysfunction (EF < 25% on echo)
* short life expectacy (below < 1 year)
* diagnosis of cancer in the past 5 years
* diagnosis of hematological diseases
* diagnosis of severe heart disease of other etiologies including valvular heart disease, Chagas' disease, etc)
* diagnosis of acute coronary syndrome in the past 3 months
* diagnosis of chronic kidney disease stage V requiring chronic dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Increase in myocardial perfusion | 1, 6 and 12 months
  Patients will undergo myocardial perfusion assessment by MRI during pharmacological stress with adenosine or dipyridamole. Alternatively, cardiac scintigraphy can be used in patients with contra-indications to MRI.

SECONDARY OUTCOMES:
Improvement in LV function | 1, 6 and 12 months
  LV function (global and regional) will be assessed by MRI.

OTHER OUTCOMES:
Improvement in angina functional class | 1, 6 and 12 months
  Angina functional class will be determined using the Canadian Cardiovascular Society classification.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Eduardo Krieger, MD, PhD, Study Director — Heart Institute; Carlos Eduardo Rochitte, MD, PhD, Study Chair — Heart Institute
Locations (1):
- Heart Institute, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Tura BR, Martino HF, Gowdak LH, dos Santos RR, Dohmann HF, Krieger JE, Feitosa G, Vilas-Boas F, Oliveira SA, Silva SA, Bozza AZ, Borojevic R, de Carvalho AC. Multicenter randomized trial of cell therapy in cardiopathies - MiHeart Study. Trials. 2007 Jan 18;8:2. doi: 10.1186/1745-6215-8-2. PMID 17233910
- [Derived] Gowdak LHW, Schettert IT, Rochitte CE, de Carvalho LP, Vieira MLC, Dallan LAO, de Oliveira SA, Cesar LAM, Brito JOR, Guarita-Souza LC, de Carvalho ACC, Krieger JE. Additional improvement in regional myocardial ischemia after intracardiac injection of bone marrow cells during CABG surgery. Front Cardiovasc Med. 2023 Feb 7;10:1040188. doi: 10.3389/fcvm.2023.1040188. eCollection 2023. PMID 36824456